CLINICAL TRIAL: NCT00378495
Title: Miltefosine for Brazilian Visceral Leishmaniasis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: accrual criteria being reviewed
Sponsor: AB Foundation (Other)
Collaborators: AEterna Zentaris (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D-18506-Z019
Record Dates: First submitted 2006-09-18; First posted 2006-09-20 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2011-01

CONDITIONS: Kala Azar
Keywords: miltefosine; kala azar; Brazil
MeSH Terms: conditions — Leishmaniasis, Visceral

INTERVENTIONS:
Drug: Miltefosine: initially 2.5 mg/kg/day for 28 days

SUMMARY:
Miltefosine will be administered to Brazilian patients with kala azar

DETAILED DESCRIPTION:
Miltefosine will be administered to Brazilian patients with kala azar. Both pediatric and adult patients will be studied. Patients will be followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed (untreated) visceral leishmaniasis with symptomatic disease and visualization of amastigotes in tissue samples or a positive culture.

  * Age: Group 1: 2 to 12 years; Group 2: 13 to 60 years
  * Sex: male and female patients eligible (no effort to be made to balance the study for gender)

Exclusion Criteria:

Exclusion criteria

Safety concerns:

* Thrombocyte count <30 x 109/l;
* Leukocyte count <1 x 109/l;
* Hemoglobin <5 g/100 ml;
* ASAT, ALAT, AP >3 times upper limit of normal range;
* Serum creatinine or BUN >1.5 times upper limit of normal range;
* Evidence of serious underlying disease (cardiac, renal, hepatic or pulmonary);
* Immunodeficiency or antibody to HIV;
* Severe protein and/or caloric malnutrition (Kwashiorkor, Marasmus);
* Any non-compensated or uncontrolled condition;
* Lactation, pregnancy (to be determined by adequate test) or inadequate contraception in females of childbearing potential for treatment period plus 2 months.

Lack of suitability for the trial:

* Negative bone marrow aspirate (smear);
* Any history of prior anti-leishmania therapy;
* Any condition which compromises ability to comply with the study procedures;
* Concomitant serious infection other than visceral leishmaniasis (this would include evidence of other conditions associated with splenomegaly such as schistosomiasis or malaria).

Administrative reasons:

* Lack of ability or willingness to give informed consent (patient and/or parent / legal representative);
* Anticipated non-availability for study visits/procedures.

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2005-04; Primary Completion 2007-04 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
cure rate at 6 months

SECONDARY OUTCOMES:
cure rate at 1 month
safety

CONTACTS AND LOCATIONS:
Overall Officials: Reynaldo Dietze, Principal Investigator — Núcleo de Doenças Infecciosas - UFES
Locations (1):
- Universidade Estadual de Montes Claros, Montes Claros, Brazil